CLINICAL TRIAL: NCT04594954
Title: Effects of Fecal Microbiota Transplantation on Weight in Obese Patients With Non-alcoholic Fatty Liver Disease: A Pilot Randomized Controlled Trial
Brief Title: Effects of Fecal Microbiota Transplantation on Weight in Obese Patients With Non-alcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-FMT-01
Record Dates: First submitted 2020-09-14; First posted 2020-10-20 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet + Exercise + FMT (Experimental)
  Interventions: Dietary Supplement: Diet; Other: FMT; Other: Physical Activity
- Diet+Exercise (Active Comparator)
  Interventions: Dietary Supplement: Diet; Other: Physical Activity

INTERVENTIONS:
Dietary Supplement: Diet — A high-protein low carbohydrate diet (HPLC) diet would be prescribed to the patients. HPLC (high-protein low carbohydrate) diet would comprise of energy as 20-25 Kcal/Kg IBW/day (amounting to 700- 800 Kcal less than the usual dietary intake), Protein as 1.2-1.5 gm/Kg IBW/day i.e. 30% of the total calories as proteins, 52% of carbohydrates 18% of fats with dietary fiber as 25 g/day. The protein requirements would be met with modular high protein, low calorie supplements.
Other: FMT — Stool Administration Procedure (ILBS FMT Protocol)
  * 500 mL filtrates will be delivered through the UGI Endoscopy into proximal jejunum [(2 to 3 minutes per 50 ml).]
  * The recipient will be kept nil per oral for at least 4 hours prior to the stool instillation.
  * 100 mL freshly thawed sample will be given once in 15 days for 3 doses
  * Non-absorbable antibiotics will be avoided in the patient from the time of enrollment into the study and therapy initiation.
  * Intravenous antibiotics will be continued as per institutional protocol in the event of active sepsis based on culture and sensitivity.
  * The patient will be allowed to consume liquid diet two hours after the procedure.
  Arms: Diet + Exercise + FMT
Other: Physical Activity — Physical Activity:
  The exercise program would consist of brisk walking. Brisk walking is defined as the walking intensity of 60-70% of their respective age-predicted maximum heart rate (target heart rate) 27,28. Speed of 5- 6 kmph considered as a brisk walking in most of the studies preferably on a treadmill for a duration of 30-45 minutes30 or brisk walking (walking faster than normal pace, measure 5000 steps continuously by pedometer). Same amount of physical activity would be prescribed to both the groups for 5 days a week for 30 -45 min.

SUMMARY:
The worldwide impact of obesity suggests an urgent need for solutions to decrease its burden on modern society. It has been generally understood that obesity is caused by a simple imbalance in the intake of energy in the form of food compared with the expenditure of energy by the body the human microbiota consists of a wide variety of microorganisms, including bacteria, archaea, fungi, viruses, protozoans and yeast. These organisms colonize both the exterior and interior of the human body in numbers that are equivalent to those of human cells of their host. Current research has identified numerous physiological and psycho-modulatory functions of the gut microbiota, including digesting food, stimulating cell growth, strengthening the immune system, preventing allergies and diseases, and impacting emotion. The gut microbiota can contribute to host physiology through metabolite production, such as short-chain fatty acids (SCFAs), which can modulate the intestinal barrier and inflammation 9.Dysbiosis of the gut microbiota, defined as a decrease in commensal bacteria levels and diversity, has been linked to diseases such as stomach/colon/liver cancer 2, obesity 9,inflammatory bowel disease (IBD) and anxiety.

DETAILED DESCRIPTION:
Aim &Objectives.

Hypothesis • Null Hypothesis: There is no difference between the Lean donor Faecal microbiota transplantation and no Faecal microbiota transplantation as regards to weight loss in obese persons with Non-alcoholic fatty liver disease

• Alternate hypothesis: Lean donor Faecal microbiota transplantation will lead to greater weight loss in obese persons with Non-alcoholic fatty liver disease as compared to no faecal microbiota transplantation in obese persons with Non-alcoholic fatty liver disease

AIM: Effects of Fecal Microbiota Transplantation on Weight in Obese Patients with Non-Alcoholic Fatty Liver Disease: A Pilot Randomized Controlled Trial.

FMT Technique:

Stool Donor Criteria A healthy single donor will be identified who will be the universal donor for all patients enrolled in the study.

The donor will be screened for

* Routine laboratory tests
* Hemogram
* Fasting blood sugar
* Liver function tests
* Lipid profile
* Stool routine and microscopy for ova & cyst, stool culture, Clostridium difficile toxin; Helicobacter pylori stool antigen; Cryptosporidium &Isospora (acid fast stain); Rotavirus antigen.
* HBsAg
* Anti-HCV
* HIV 1 & 2
* VDRL
* HLA A1
* BMI is between 18- 21 and waist circumference < 90 cm in men and < 80 cm in women (all 3 fulfilled).

Donor will be excluded if he/she has:

* Abnormal bowel motions
* Chronic alcohol intake
* Active substance abuse or failed to provide consent
* Less than 18 or more than 60 years of age
* HBsAg, Anti HCV, HIV seropositivity
* Gastroenteritis within last 2 months
* Inflammatory bowel disease
* Any malignancy
* Chronic kidney disease, coronary artery disease, CVA, COPD, DM-2
* Antibiotic usage within 3 months at the time of enrolment.
* Transaminitis, dyslipidemia, Ova/ Cyst in stools, Clostridium deficile toxin+

Stool donor procedure:

* Donor will be advised to follow a normal diet plan during the study process, in consultation with the hospital dietician.
* Donor will not be permitted to eat street foods or to eat at public/family functions or parties from the time of enrollment till completion of protocol.

Stool Collection and Preparation:

* Donor will be advised to collect and submit fresh stool sample on the day of the planned procedure.
* Stool specimen (preferably Bristol Stool Type 4 or 5) with a weight of ∼250 g will be considered adequate.
* 250gm stool sample form the selected donor will be resuspended in 250ml of freezing media. This will be agitated in a blender 3 times in pluses of 20-30seconds to get a homogenate. The freezing media will contain 12.5% glycerol and 0.9% N saline.
* The homogenous suspension will then be filtered through sterile gauze pieces, 3-4 times.
* 30ml filtrate will be collected in aliquot of 100 ml volume and this will be stored at -80C till use.
* For use the aliquot containing 30ml of filtrate will be thawed at 30C in a warm water bath. 70ml 0.9%N saline will be added to make up the volume to 100ml.

Stool Administration Procedure (ILBS FMT Protocol)

* 500 mL filtrates will be delivered through the UGI Endoscopy into proximal jejunum [(2 to 3 minutes per 50 ml).]
* The recipient will be kept nil per oral for at least 4 hours prior to the stool instillation.
* 100 mL freshly thawed sample will be given once in 15 days for 3 doses
* Non-absorbable antibiotics will be avoided in the patient from the time of enrollment into the study and therapy initiation.
* Intravenous antibiotics will be continued as per institutional protocol in the event of active sepsis based on culture and sensitivity.
* The patient will be allowed to consume liquid diet two hours after the procedure.

Post-Procedure Advice and Management

* Rifaximin, LAXATIVES and other non-absorbable antibiotics will be withheld.
* Antibiotics will be given in both the groups when clinically indicated.

DIET AND EXERCISE PROGRAMME AND ASSESSMENT OF COMPLIANCE:

Dietary Intervention:

A high-protein low carbohydrate diet (HPLC) diet would be prescribed to the patients. HPLC (high-protein low carbohydrate) diet would comprise of energy as 20-25 Kcal/Kg IBW/day (amounting to 700- 800 Kcal less than the usual dietary intake), Protein as 1.2-1.5 gm/Kg IBW/day i.e. 30% of the total calories as proteins, 52% of carbohydrates 18% of fats with dietary fiber as 25 g/day. The protein requirements would be met with modular high protein, low calorie supplements25,26.

Physical Activity:

The exercise program would consist of brisk walking. Brisk walking is defined as the walking intensity of 60-70% of their respective age-predicted maximum heart rate (target heart rate) 27,28. Speed of 5- 6 kmph considered as a brisk walking in most of the studies preferably on a treadmill for a duration of 30-45 minutes30 or brisk walking (walking faster than normal pace, measure 5000 steps continuously by pedometer). Same amount of physical activity would be prescribed to both the groups for 5 days a week for 30 -45 min

Duration of Intervention: This diet and exercise regimen would be implemented for a period of 6months

Assessment of Compliance- Following measures would be taken to ensure the compliance of the patients-

1. Diet Charts: - Individual diet charts (customized to patient's requirements) - mentioning the total amount of food items, their quantity & house hold measure would be provided and explained, for a lucid understanding.
2. Daily diet dairy: - All the patients would record their daily diet in a dairy given to them, to maximize their adherence and self-motivation to comply with the prescribed diet.
3. Telephonic follow-ups: - Weekly, all the patients would be telephoned to check their overall compliance with the prescribed diet.
4. Follow-up in OPD: - Patient would be asked to follow-up in the OPD at 1 month to check their overall clinical progress and compliance. The diet and symptom diary would be cross checked and also confirmed with the nearest relative.
5. The overall compliance: - The compliance questionnaire is one of the methods to ensure compliance (other than diet charts, diet diary, OPD follow-ups and telephonic follow-ups) and an objective way to quantify the overall dietary compliance of the patients. In point number 5 the calculation of the Likert scale (3 options) is very explicitly given, nevertheless the actual questionnaire is a modified version of the one used in the study of the Abdullah Al Lahiri's paper. This modified questionnaire is attached in the Performa. Likert scale based questionnaire24, including 10 close-ended questions. Responses would be rated on a three-point scale, which would be required to determine whether the patients (always=2, sometimes=1 or never=0) followed dietary advice. According to the overall score, which would range from 0 to 20, the patient's adherence would be classified as- i. 'Good adherence' if the score is >15 ii. 'Partial adherence' if the score is between 10 and 15 iii. 'Non-adherence' if the score is <10.

Amount of food is going to based upon each individual. We will give diet chart to every individual; we will explain to each individual in details regarding the benefits of protein low carbohydrate and the importance of the quantification of the diet. Regarding the scale of compliance, it is validated and used also and I have attached the questionnaires in the Performa. Exemplary diet chart also attached in the Performa.

Physical activity compliance: -

1. First Session at study facility: Patient will be asked to complete one session of the prescribed exercise at the study facility so that they understand the regimen well and can do the rest at home.
2. Activity log book: Patients will be asked to fill the activity log books on daily basis and bring it every time they visit the OPD.
3. It is measured by self-report questionnaires. There are so many self-report questionnaires like Modifiable Activity Questionnaire (MAQ), Previous Week Modifiable Activity Questionnaire (PWMAQ), Recent Physical Activity Questionnaire (RPAQ), International Physical Activity Questionnaires (IPAQ), Previous Day Physical Activity Recall (PDPAR), and 7-day Physical Activity Recall (PAR) 31,. International Physical Activity Questionnaire (IPAQ) - Short Form: IPAQ-SF will be used at baseline and at the end of the intervention period to assess the type of physical activity and sitting time. Total physical activity is expressed in MET-min/week and time spent in sitting will be calculated during the last 7 days. According to the MET-min/week physical activity level of the patients would be categorized as Vigorous, Moderate or Low. Likewise changes in the MET-min/week would express not only the compliance of the patient but also take into account the any additional activities done by the patient other than the minimum prescribed ones Donor diet during FMT The selected donor is a single healthy lean young person, having a desired body weight. Hence during the study period (i.e. till the donor is donating the stool sample in the study) the donor would be asked to follow his usual normal diet and there would not be any specifications for the 'type' of diet he is supposed to eat. Nevertheless, in order to avoid any eventualities of gastrointestinal disorders which would necessitate use of antibiotics and other drugs hampering the stool donation process, this healthy donor would be asked to abstain from eating street foods. However, he is free to eat at family get-togethers and parties, if any.

FOLLOW-UP OF PATIENTS [AT BASELINE, 3 MO, 6 MO AND 12 MO].

Life style failure is defined as Dietary therapy should ensure an intake reduced by 500 to 1,000 kcal/day from the current level. Low calorie diets (LCDs) containing 1,000 to 1,200 kcal/day for most women and between 1,200 kcal/day and 1,600 kcal/day for men. Physical activity (walking, dancing, gardening, household chores and team or individual sports) should be increased slowly to a level that ensures at least 30 minutes or more of moderate-intensity physical activity on most, and preferably all, days of the week for 6 months could not reduce weight by 5 % labeled as life style failure.

Body Weight: - electronic weighing machine.

Waist and Hip Measurements :- the waist circumference should be measured at the midpoint between the lower margin of the last palpable ribs and the top of the iliac crest, using a stretch-resistant tape that provides a constant 100 g tension. Hip circumference should be measured around the widest portion of the buttocks, with the tape parallel to the floor. 14

Clinical Laboratory Assessments. Insulin resistance (HOMA-IR): - (Insulin resistance (HOMA-IR): - fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.) and insulin is getting measured by A chemiluminescent immunoassay (CLIA) 15 is commonly used in our laboratories for measurement of insulin concentration in our samples.

High-sensitivity C-reactive protein, fibrinogen TNF-alpha, adiponectin, leptin, Ghrelin.: - they are measured with the special ELISA kit.

Gut microbiome analysis methods: - This technique allows the rapid sequencing of multiple samples at one time, yielding thousands of sequences reads per sample. Specifically, we generated a set of 96 emulsion polymerase chain reaction (PCR) fusion primers that contain the 454 emulsion PCR linkers on the 27F primer (AGAGTTTGATCCTGGCTCAG-3=) and 355R' (5=-GCTGCCTCCCGTAGGAGT-3=) and different 8-base barcode between the A adapter and the 27F primer.8 Thus, each faecal sample was amplified with unique bar-coded forward 16S ribosomal RNA primers, and then up to 96 samples were pooled and subjected to emulsion PCR and pyro sequenced. 16

Serum transcriptome: - Transcriptomics technologies are the techniques used to study an organism's transcriptome, the sum of all of its RNA transcripts. The information content of an organism is recorded in the DNA of its genome and expressed through transcription. Here, mRNA serves as a transient intermediary molecule in the information network, whilst noncoding RNAs perform additional diverse functions. A transcriptome captures a snapshot in time of the total transcripts present in a cell. The first attempts to study the whole transcriptome began in the early 1990s, and technological advances since the late 1990s have made transcriptomics a widespread discipline. Transcriptomics has been defined by repeated technological innovations that transform the field. There are two key contemporary techniques in the field: microarrays, which quantify a set of predetermined sequences, and RNA sequencing (RNA-Seq), which uses high throughput sequencing to capture all sequences. 17

Body composition analysis method: - common assessments are anthropometric and include weight, stature, abdominal circumference, and skinfold measurements. 18 Assessment of compliance to diet and exercise programme: - by the number of questionnaires asked during each visit of patient in the hospital.

Stool sample for microbiome analysis will be collected on day 0,7, 90 and 180. All the adverse effects will be monitored and notified.

Study population: 18- 55 yrs of age with NAFLD and

* BMI ≤ 35 or
* Body Mass Index (BMI) is ≤30 to 34.9 kg/m2 with at least one treated or untreated comorbid condition (hypertension, dyslipidaemia, cardiovascular disease, glucose intolerance, sleep apnoea, NASH).

Attended hepatology OPD. Study design: Randomized controlled trial Study period: One year from ethics approval. Sample size: 110 (55 cases in each group) Intervention: The subjects will be given FMT through UGI endoscopy. They will be administered the processed fecal microbiota sample collected from lean healthy donor for a period of 0/15/30 days.

FOLLOW-UP OF PATIENTS [AT BASELINE, 3 MO, 6 MO AND 12 MO]

* Body Weight
* Waist and Hip Measurements
* Clinical Laboratory Assessments
* Insulin resistance (HOMA-IR) (Insulin resistance (HOMA-IR): - fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.)
* High-sensitivity C-reactive protein, fibrinogen TNF-alpha, adiponectin, leptin, Gherlin.
* Gut microbiome analysis
* Serum transcriptome
* Body composition analysis Assessment of compliance to diet and exercise programme
* Stool sample for microbiome analysis will be collected on day 0,7, 90 and 180, 360
* All the adverse effects will be monitored and notified. Monitoring and assessment: -all the parameters of the objective and also noted any adverse effects.

Adverse effects: diarrhea, pneumonia, abdominal pain, constipation, nausea vomiting, fever and death Stopping rule: In the event of any of the adverse effects during therapy.

Ethical issues in the study and plans to address these issues: None

ELIGIBILITY:
Inclusion Criteria:

1. Patients posted for Upper GI endoscopy for other indications
2. 18- 55 yrs of age with NAFLD and
3. BMI ≤ 35 or
4. Body Mass Index (BMI) is ≤30 to 34.9 kg/m2 with at least one treated or untreated comorbid condition (hypertension, dyslipidaemia, cardiovascular disease, glucose intolerance, sleep apnoea, NASH).
5. Ambulatory and able to perform the ILBS healthy lifestyle (diet and exercise program).
6. Failed to life style therapy.

Exclusion Criteria:

1. HIV, HBsAg or HCV positive
2. Prior bariatric surgery
3. Change in weight of ≤5 % within 3 months
4. Malignancy within 5 years
5. Recent major surgery; history of seizure disorder
6. Depression or other major psychiatric disease within 2 years requiring treatment with prescription medication
7. Pregnancy or lactation
8. Significant uncontrolled cardiopulmonary diseases
9. Major surgical procedure (intrathoracic, intracranial, intraperitoneal, liposuction) within 6 months of screening
10. Hypo or hyperthyroidism uncontrolled. If initiation or adjustment of doses of these drugs is anticipated, patients should not be enrolled.
11. Patients being treated for hypothyroidism must be adequately replaced on a stable dose of medication for at least 3 months prior to screening.
12. Uncontrolled DM with HbA1c greater than 9%.
13. Recent treatment (i.e., within 1 month of the screening visit) with weight drugs or products or appetite suppressants (including herbal weight agents)
14. Recent treatment (i.e., within 3 months of the screening visit) with oral or parenteral corticosteroids
15. Recent history (within 2 years prior to the screening visit) of significant alcohol use
16. Significant change in diet or level of physical activity within 1 month prior to enrolment
17. Use of very-low calorie (< 1,000/day) liquid weight diet within 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving ≤ 5%of the weight loss in kg from baseline | 3 months

SECONDARY OUTCOMES:
Proportion of patients achieving ≤ 5% of the weight loss in kg from baseline | 6 months
Proportion of patients achieving ≤ 5% of the weight loss in kg from baseline | 12 months
Changes in waist circumference and waist hip ratio | 3 months
Changes in waist circumference and waist hip ratio | 6 months
Changes in waist circumference and waist hip ratio | 1 year
Changes in systolic and diastolic BP | 3 months
Changes in systolic and diastolic BP | 6 months
Changes in systolic and diastolic BP | 1 year
Changes in Total cholesterol in both groups | 3 months
Changes in Total cholesterol in both groups | 6 months
Changes in Total cholesterol in both groups | 1 yera
Changes in LDL cholesterol in both groups | 3 months
Changes in LDL cholesterol in both groups | 6 months
Changes in LDL cholesterol in both groups | 1 year
Changes in Triglyceride levels in both groups | 3 months
Changes in Triglyceride levels in both groups | 6 months
Changes in Triglyceride levels in both groups | 1 year
Changes in Fasting glucose in both groups | 3 months
Changes in Fasting glucose in both groups | 6 months
Changes in Fasting glucose in both groups | 1 year
Changes in insulin in both groups | 3 months
Changes in insulin in both groups | 6 months
Changes in insulin in both groups | 1 year
Changes in HbA1C in both groups | 3
Changes in HbA1C in both groups | 6 months
Changes in HbA1C in both groups | 1 year
Changes in homeostasis model assessment of insulin resistance in both groups | 3 months
Changes in homeostasis model assessment of insulin resistance in both groups | 6 months
Changes in homeostasis model assessment of insulin resistance in both groups | 1 year
Changes in fibroscan values in both groups | 6 months
Changes in fibroscan values in both groups | 12 months
Changes in CAP values in both groups | 6 months
Changes in CAP values in both groups | 12 months
Changes in High-sensitivity C-reactive protein in both groups | 3 months
Changes in High-sensitivity C-reactive protein in both groups | 6 months
Changes in High-sensitivity C-reactive protein in both groups | 1 year
Change in Fibrinogen in both groups | 3 months
Change in Fibrinogen in both groups | 6 months
Change in Fibrinogen in both groups | 12 months
Change in TNF alpha in both groups | 3 months
Change in TNF alpha in both groups | 6 months
Change in TNF alpha in both groups | 12 months
Changes in faecal microbiome in both groups | 3 months
Changes in faecal microbiome in both groups | 6 months
Changes in faecal microbiome in both groups | 1 year
Changes in body composition in both groups | 3 months
  Body composition will be done by Body Composition Analysis Machine
Changes in body composition in both groups | 6 monhs
  Body composition will be done by Body Composition Analysis Machine
Changes in body composition in both groups | 1 year
  Body composition will be done by Body Composition Analysis Machine
Changes in quality of life in both groups | 3 months
Changes in quality of life in both groups | 6 months
Changes in quality of life in both groups | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided